CLINICAL TRIAL: NCT04447248
Title: Quantitative Cardiotocography and Doppler Ultrasound in the Detection of Hypoxia Among Growth-restricted Fetuses
Brief Title: qCTG and Doppler Ultrasound in the Detection of Hypoxia Among FGR Fetuses
Status: Completed | Type: Observational
Sponsor: Orthogyn Medical Center, Bulgaria (Other)
Responsible Party: Principal Investigator, Petar Ignatov, Assist. Prof. Petar Ignatov, MD, Ph.D., Orthogyn Medical Center, Bulgaria
Other Study IDs: QDSP Protocol
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Late-onset Fetal Growth Restriction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: QDSP Protocol — Computerized expert system for fetal monitoring, based on cardiotocogrpaphy

SUMMARY:
To evaluate the benefits of combining Doppler measurements of placental/fetal blood vessels with computerized cardiotocography (quantitative cardiotocogrpahy - qCTG) in the detection of fetal hypoxia (pH < 7.20) among late-onset growth restricted (SGR) fetuses

ELIGIBILITY:
Inclusion Criteria:

* estimated fetal weight below the 10th centile of the reference curve for the Bulgarian population (11);
* absence of sonographic and laboratory evidence of structural anomalies;
* absence of severe maternal complications;
* documented birth weight < 10th centile;
* full follow-up documentation

Exclusion Criteria:

* multiple pregnancies;
* congenital malformations and any chromosomal malformations known before labor and delivery;
* severe maternal complications;
* documented birth weight > 10th centile;
* pregnancy loss;
* failure to obtain full follow-up documentation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Bulgarian population (caucasian)
Sampling Method: Non-Probability Sample
Enrollment: 1714 (Actual)
Dates: Start 2011-05-05 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Occurence of hypoxia (pH<7.20) at birth | up to 5 minutes after delivery

IPD SHARING:
Plan to Share IPD: Undecided